CLINICAL TRIAL: NCT00002310
Title: A Pilot Study to Determine the Safety and Efficacy of Topically Applied SP-303T in Patients With Acquired Immunodeficiency Syndrome and Concomitant Herpes Simplex Virus (HSV) Infection Unresponsive to Acyclovir
Brief Title: SP-303T Applied to the Skin of Patients With Herpes Simplex Virus (HSV) Infection and AIDS Who Have Not Had Success With Acyclovir
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaman Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 120A; SP303T-A-01
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1993-09

CONDITIONS: Herpes Simplex; HIV Infections
Keywords: Herpes Simplex; HIV-1; Acquired Immunodeficiency Syndrome; Antiviral Agents; Administration, Topical
MeSH Terms: conditions — Herpes Simplex; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — crofelemer

INTERVENTIONS:
Drug: Crofelemer

SUMMARY:
To evaluate the safety and tolerance of topically applied SP-303T in AIDS patients. To observe the effect of this drug on herpes simplex virus lesions in patients who have failed to heal in response to oral or intravenous acyclovir therapy.

The lack of alternative treatments for herpes simplex virus infection in patients with AIDS and the development of resistance to acyclovir for patients requiring repeated treatment presents a therapeutic dilemma for physicians. SP-303T has good in vitro activity against resistant strains and offers a convenient and inexpensive means of drug administration in comparison to the use of intravenous medication.

DETAILED DESCRIPTION:
The lack of alternative treatments for herpes simplex virus infection in patients with AIDS and the development of resistance to acyclovir for patients requiring repeated treatment presents a therapeutic dilemma for physicians. SP-303T has good in vitro activity against resistant strains and offers a convenient and inexpensive means of drug administration in comparison to the use of intravenous medication.

Patients receive 14 days (and up to 42 days) of treatment with topically applied SP-303T. SP-303T is applied directly onto herpes simplex virus lesions three times daily in a quantity sufficient to thinly cover the entire lesion, which may then be covered with an appropriate dressing, if needed. At the end of the treatment period, patients enter a follow-up period of 2 weeks.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV-1 infection.
* AIDS.
* Chronic mucocutaneous herpes simplex virus (HSV) infection, with one or more lesions unresponsive to oral acyclovir therapy.
* No uncontrolled infections other than HSV.
* Sufficient mental status to understand the purpose of the study and to comply with study requirements.
* Sufficient general health to be an outpatient and to come to the clinic for required follow-up visits.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Known hypersensitivity or allergy to citrus fruits, black currant berries, and rose hips.
* Any disease condition that, in the opinion of the investigator, would interfere with evaluation of the study drug, affect patient compliance, or place the patient at increased risk.

Concurrent Medication:

Excluded:

* Other unapproved investigational new drugs.
* Concurrent other therapy for herpes simplex virus (HSV) infection or medications with known activity against HSV.

Required:

* A minimum of 10 days of prior oral acyclovir (at least 1 g daily) or 10 days of prior intravenous acyclovir (15 mg/kg daily).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - UCSF - San Francisco Gen Hosp, San Francisco, California
  - TheraFirst Med Ctrs Inc, Fort Lauderdale, Florida
  - Saint Luke's - Roosevelt Hosp Ctr, New York, New York
  - Univ of Utah School of Medicine, Salt Lake City, Utah